CLINICAL TRIAL: NCT00083902
Title: UARK 98-025, A Randomized Phase II Trial of Dexamethasone or Dexamethasone in Combination With Thalidomide as Salvage Therapy for Low-Risk Post Transplantation Relapse in Patients With Multiple Myeloma
Brief Title: Dexamethasone or Dexamethasone in Combination With Thalidomide as Salvage Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UARK 98-025
Record Dates: First submitted 2004-06-03; First posted 2004-06-04 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-07

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Thalidomide; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Thalidomide; Dexamethasone

INTERVENTIONS:
Drug: Thalidomide
Drug: Dexamethasone

SUMMARY:
The purpose of this investigational trial is to find out how well patients respond and how long their response lasts when treated with a standard regimen of dexamethasone with or without thalidomide and also find out what kind of side effects patients will experience.

DETAILED DESCRIPTION:
Maintenance

Dexamethasone

Patients will receive 40 mg dexamethasone days 1-4 only, every 3-4 weeks. Response will be assessed at least every 3 months while on maintenance therapy. Appropriate H2 blocker and antibiotics will also be given.

Thalidomide

Thalidomide will continue at a dose of 400 mg daily, or at the dose that was reduced and judged to be well tolerated in induction therapy. Thalidomide will be given as an oral, once daily dose at bedtime. Those patients unable to tolerate dexamethasone may continue on thalidomide alone until criteria for removal from treatment is met.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a confirmed diagnosis of previously treated, active multiple myeloma, with hypoproliferative/low risk relapse following at least one autologous transplant.
* Patients must be 18 years of age or older. Women of childbearing age and fertile men must use a medically acceptable means of birth control while on study and for 6 months thereafter.
* Patients must sign an informed consent to participate in this study, and be fully aware of the known teratogenic potential of this drug combination.
* Patients must have a SWOG performance status of 0-2.
* Patients must have adequate renal function, as defined by serum creatinine < or = 3.0 mg/dl.
* Patients must be off chemotherapy (including steroids) and local radiotherapy for > or equal 3 weeks prior to entering the study.

Exclusion Criteria:

* No other concurrent therapy for myeloma is permitted while on protocol.
* There must be no evidence of active infection requiring IV antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190
Dates: Start 1998-06; Study Completion 2005-05

PRIMARY OUTCOMES:
To evaluate the effectiveness of dexamethasone (dex) alone as compared to dex in combination with thalidomide in low risk patients relapsing after autologous transplantation.

SECONDARY OUTCOMES:
To evaluate the quantitative and qualitative toxicities associated with the regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Zangari, M.D., Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States

REFERENCES:
- See also: Myeloma Institute for Research & Therapy website — http://myeloma.uams.edu